CLINICAL TRIAL: NCT03949803
Title: Effect of the Timing of Chocolate Intake on Body Fat Distribution, Substrate Oxidation, and Microbiota. Randomized, Crossover Study
Brief Title: Eating Chocolate at the Right Time Benefits the Circadiam Sytem and Metabolic Efficiency.
Acronym: ONTIME-CHOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Murcia (Other)
Responsible Party: Principal Investigator, PROF. MARTA GARAULET AZA, Principal Investigator, Universidad de Murcia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2017ES00004
Record Dates: First submitted 2018-02-08; First posted 2019-05-14 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Menopause
Keywords: Chocolate; Timing; Menopause; Calorimetry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Morning Chocolate, then Evening/Night Chocolate and Control Chocolate (Experimental): First condition is eating 100gr chocolate within one hour of habitual waketime. Second condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Third condition is eating no milk chocolate or other chocolate.
  Interventions: Behavioral: Chocolate 100gr
- Morning Chocolate, then Control Chocolate and Evening/Night Chocolate (Experimental): First condition is eating 100gr chocolate within one hour of habitual waketime. Second condition is eating no milk chocolate or other chocolate. Third condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Interventions: Behavioral: Chocolate 100gr
- Evening/Night Chocolate, then Morning Chocolate and Control Chocolate (Experimental): First condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Second condition is eating 100gr chocolate within one hour of habitual waketime.
  Third condition is eating no milk chocolate or other chocolate.
  Interventions: Behavioral: Chocolate 100gr
- Evening/Night Chocolate, then Control Chocolate and Morning Chocolate (Experimental): First condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Second condition is eating no milk chocolate or other chocolate. Third condition is eating 100gr chocolate within one hour of habitual waketime.
  Interventions: Behavioral: Chocolate 100gr
- Control Chocolate, then Morning Chocolate and Evening/Night Chocolate (Experimental): First condition is eating no milk chocolate or other chocolate. Second condition is eating 100gr chocolate within one hour of habitual waketime.
  Third condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Interventions: Behavioral: Chocolate 100gr
- Control Chocolate, then Evening/Night Chocolate and Morning Chocolate (Experimental): First condition is eating no milk chocolate or other chocolate. Second condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime.
  Third condition is eating 100gr chocolate within one hour of habitual waketime.
  Interventions: Behavioral: Chocolate 100gr

INTERVENTIONS:
Behavioral: Chocolate 100gr — Evening/Night Chocolate:
  Eating 100gr of milk chocolate within 1 hours of habitual bedtime
  Control Chocolate:
  Eating no milk chocolate or other chocolate
  Chocolate Morning:
  Eating chocolate within one hour of habitual waketime.

SUMMARY:
The purpose of this investigation is to test the hypothesis that in humans, eating a relatively big amount of chocolate at the wrong time (bedtime) may disrupt our circadian system (change the circadian phase), while taking this same amount of chocolate in the morning (wake up condition) may synchronize it. Other related factors may be also affected such as total body weight and body fat, dietary habits (total energy intake and macronutrient distribution), the timing of food intake and of sleep, daily rhythms of TAP, microflora composition and postprandial glycemia.

DETAILED DESCRIPTION:
Recent studies suggest that not only "what" the people eat, but also "when" the people eat may have a significant role in obesity treatment and in the regulation of the circadian system. Thus, the hypothesis of this study is eating a relatively big amount of chocolate at the wrong time, bedtime may affect:

1. Metabolism: resting energy expenditure, corrected resting energy respiratory quotient (RQ)
2. Glucose metabolism
3. Total weight loss
4. Food intake, total energy intake, and type of food
5. Microflora (feces)
6. Mood
7. Disrupt our circadian system 7a) Changes in Temperature, Actimetry, and Position 7b) Electrocardiogram (ECG) 7c) Melatonin (two points) cortisol rhythm (three points) While having this same amount of chocolate in the morning (wake up condition) may synchronize it.

Other related factors may be also affected such as total body weight and body fat, dietary habits (total energy intake and macronutrient distribution), the timing of food intake and of sleep, daily rhythms of TAP, microflora composition and postprandial glycemia.

19 women (postmenopausal) following the habitual dietary habits of participants (ad libitum) will have 30% of the habitual total daily calories in chocolate of participants (Nestle, "chocolate with milk") during two consecutive weeks each under three conditions: eating chocolate within 1 hour of habitual wake-time, eating chocolate within 1 hours of habitual bedtime, or eating no chocolate. No other chocolate (i.e., none at all in control and in the washout weeks).

The protocol will be a randomized, cross-over design, with a 1-week washout between each condition.

During the 14 days in each condition, the participants will record sleep and activity schedules by dairy, food intake and food timing by phone application, daily rhythms of wrist temperature, activity and position (TAP).

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Age: between 45 and 65 year of age
* Caucasian
* Menopause

Exclusion Criteria:

* Pre-menopause women
* Endocrine (Diabetes mellitus or others), renal, hepatic, cancer or psychiatric disorders
* Receiving any pharmacologic treatment other than oral contraceptives
* Bulimia diagnosis, prone to binge eating
* Pregnancy

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-01-15 (Actual); Study Completion 2017-04-20 (Actual)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hernandez-Gonzalez T, Gonzalez-Barrio R, Escobar C, Madrid JA, Periago MJ, Collado MC, Scheer FAJL, Garaulet M. Timing of chocolate intake affects hunger, substrate oxidation, and microbiota: A randomized controlled trial. FASEB J. 2021 Jul;35(7):e21649. doi: 10.1096/fj.202002770RR. PMID 34164846

RESULTS

PARTICIPANT FLOW:
Groups:
- Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate: First condition is eating 100gr chocolate within one hour of habitual waketime. Second condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime Third condition is eating no milk chocolate or other chocolate
- Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate: First condition is eating 100gr chocolate within one hour of habitual waketime. Second condition is eating no milk chocolate or other chocolate Third condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime
- Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate: First condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime Second condition is eating 100gr chocolate within one hour of habitual waketime.
  Third condition is eating no milk chocolate or other chocolate
- Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate: First condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime Second condition is eating no milk chocolate or other chocolate Third condition is eating 100gr chocolate within one hour of habitual waketime.
- Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate: First condition is eating no milk chocolate or other chocolate Second condition is eating 100gr chocolate within one hour of habitual waketime.
  Third condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime
- Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate: First condition is eating no milk chocolate or other chocolate Second condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime Third condition is eating 100gr chocolate within one hour of habitual waketime.
Period: First Intervention (2 Weeks)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Started | 3 | 3 | 5 | 2 | 3 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washsout (1 Week)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Started | 3 | 3 | 5 | 2 | 3 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (2 Weeks)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Started | 3 | 3 | 5 | 2 | 3 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washsout (1 Week)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Started | 3 | 3 | 5 | 2 | 3 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (2 Weeks)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Started | 3 | 3 | 5 | 2 | 3 | 3
Completed | 3 | 3 | 5 | 2 | 3 | 3
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate: First condition is eating 100gr of milk chocolate within 1 hours of habitual bedtime Second condition is eating 100gr chocolate within one hour of habitual waketime.
- Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate: First condition is eating no milk chocolate or other chocolate Second condition is eating 100gr chocolate within one hour of habitual waketime.
- Total: Total of all reporting groups
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate | Total
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3 | 19
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 56.00 (7.81) | 54.00 (4.58) | 50.20 (3.56) | 51.50 (9.19) | 51.00 (0.00) | 52.67 (0.58) | 52.37 (4.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 5 | 2 | 3 | 3 | 19
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Resting Energy Expenditure (Indirect Calorimetry)
Description: The investigators will measure by indirect calorimetry the resting energy expenditure after each condition (no chocolate, Morning Chocolate, Night Chocolate) Changes in Resting Energy Expenditure (Indirect Calorimetry) were determined by changes in resting energy expenditure occurred in the participants between baseline and after 2 weeks in each of the three different experimental conditions. Oxygen (O2) consumption (mL/min) and carbon dioxide (CO2) production (mL/min) were measured. The Respiratory Quotient (RQ) was calculated out of O2 consumption (mL/min) and CO2 production (mL/min). Energy expenditure values (kcal/day) were calculated according to the Weir equation: Metabolic rate (kcal per day) = 1440 (3.9 VO2 + 1.1 VCO2)*
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: kcal/day
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3
kcal/day
  Resting energy expenditure at Baseline | 1249.33 (147.56) | 1377.67 (158.80) | 1360.40 (137.06) | 1468.50 (272.23) | 1427.33 (121.71) | 1259.67 (83.29)
  Resting energy expenditure Morning Condition | 1354.33 (227.25) | 1344.00 (115.47) | 1413.80 (151.61) | 1389.00 (255.97) | 1289.67 (153.05) | 1354.00 (60.23)
  Resting energy expenditure Evening Condition | 1292.33 (126.02) | 1459.67 (30.14) | 1323.60 (174.69) | 1497.50 (208.60) | 1281.00 (187.20) | 1351.67 (60.14)
  Resting energy expenditure Control Condition | 1342.00 (45.64) | 1376.67 (95.36) | 1439.20 (175.72) | 1464.50 (27.58) | 1420.67 (69.87) | 1397.00 (105.79)

2. Primary Outcome: Total Body Weight
Description: The investigators will measure total body weight after each condition (no chocolate, Morning Chocolate, Night Chocolate)
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: kilograms (kg)
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3
kilograms (kg)
  Weight at Baseline | 64.32 (3.43) | 61.97 (8.09) | 67.87 (10.37) | 74.08 (24.50) | 64.42 (7.13) | 61.95 (14.90)
  Weight at Morning condition | 63.02 (1.76) | 62.07 (8.42) | 67.73 (10.68) | 73.35 (22.98) | 64.58 (7.28) | 63.2 (15.24)
  Weight at Night condition | 63.22 (2.28) | 62.00 (8.66) | 67.68 (10.91) | 74.25 (22.98) | 65 (6.24) | 62.67 (15.04)
  Weight at Control condition | 63.33 (2.08) | 61.00 (7.81) | 68.00 (10.49) | 74.00 (24.04) | 64.33 (7.77) | 60.67 (14.22)

3. Secondary Outcome: Fragmentation of Wrist Temperature (WT) Daily Rhythm
Description: The investigators will measure the fragmentation parameter derived from wrist temperature after each condition (no chocolate, Morning Chocolate, Night Chocolate). Intradaily variability (IV) characterizes the rhythm fragmentation.
  Changes in daily rhythm of wrist temperature fragmentation were measured by changes in the fragmentation parameter derived from wrist temperature along the two weeks of intervention in each of the three conditions. The participants wore a wristwatch during the last 7 days of each condition on the non-dominant wrist to record body temperature and activity. Wrist temperature parameters were measured to represent the wrist body temperature pattern, which provides an objectively measure of sleep and siesta (together with activity rhythm).
  A low fragmentation involves a low intraday rhythmicity of the circadian rhythm.
  Its values oscillated between 0, when the wave was perfectly sinusoidal, and 2, when the wave was as Gaussian noise.
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3
arbitrary units
  Fragmentation of WT rhythm at Baseline | 0.23 (0.11) | 0.15 (0.05) | 0.25 (0.13) | 0.18 (0.08) | 0.13 (0.05) | 0.18 (0.07)
  Fragmentation of WT rhythm at Morning condition | 0.13 (0.03) | 0.18 (0.04) | 0.15 (0.06) | 0.31 (0.06) | 0.18 (0.08) | 0.16 (0.09)
  Fragmentation of WT rhythm at Night condition | 0.15 (0.07) | 0.24 (0.09) | 0.21 (0.10) | 0.25 (0.14) | 0.17 (0.04) | 0.20 (0.14)
  Fragmentation of WT rhythm at Control condition | 0.11 (0.03) | 0.24 (0.14) | 0.12 (0.04) | 0.15 (0.04) | 0.15 (0.03) | 0.13 (0.04)

4. Secondary Outcome: Regularity of Wrist Temperature (WT) Daily Rhythm
Description: The investigators will measure the regularity parameter derived from wrist temperature after each condition (no chocolate, Morning Chocolate, Night Chocolate). RegularIty is measured as interdaily stability (IS), that means rhythm stability over different days; it varied between 0 for Gaussian noise to 1 for perfect stability, where the rhythm repeated itself exactly day after day.
  Changes in daily rhythm of wrist temperature regularity were measured by changes in the regularity parameter derived from wrist temperature along the two weeks of intervention in each of the three conditions. A regular rhythm means recurring at uniform intervals. The participants wore a wristwatch during the last 7 days of each condition on the non-dominant wrist to record body temperature and activity. Wrist temperature parameters were measured to represent the wrist body temperature pattern, which provides an objectively measure of sleep and siesta (together with activity rhythm).
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: arbitrary units
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3
arbitrary units
  Regularity of WT daily rhythm at Baseline | 0.44 (0.12) | 0.45 (0.06) | 0.49 (0.16) | 0.32 (0.04) | 0.56 (0.05) | 0.35 (0.17)
  Regularity of WT daily rhythm at Morning condition | 0.49 (0.14) | 0.43 (0.13) | 0.41 (0.07) | 0.30 (0.18) | 0.30 (0.02) | 0.44 (0.16)
  Regularity of WT daily rhythm at Night condition | 0.41 (0.22) | 0.45 (0.12) | 0.41 (0.06) | 0.40 (0.07) | 0.39 (0.20) | 0.32 (0.08)
  Regularity of WT daily rhythm at Control condition | 0.43 (0.27) | 0.34 (0.15) | 0.35 (0.05) | 0.24 (0.03) | 0.42 (0.22) | 0.29 (0.26)

5. Secondary Outcome: Amplitude of Wrist Temperature (WT) Daily Rhythm
Description: The investigators will measure the amplitude parameter derived from wrist temperature after each condition (no chocolate, Morning Chocolate, Night Chocolate). In the cosinor analysis to characterize the WT rhythm, we calculate amplitude (difference between the maximum [or minimum] value of the cosine function and mesor) Changes in daily rhythm of wrist temperature amplitude were measured by changes in the amplitude parameter derived from wrist temperature along the two weeks of intervention in each of the three conditions. The participants wore a wristwatch during the last 7 days of each condition on the non-dominant wrist to record body temperature and activity. Wrist temperature parameters were measured to represent the wrist body temperature pattern, which provides an objectively measure of sleep and siesta (together with activity rhythm).
  A healthy circadian rhythm is considered as the one with high amplitude.
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: ºC
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 2 | 3 | 3
ºC
  Amplitude of WT daily rhythm at Baseline | 0.95 (0.59) | 1.42 (0.57) | 0.92 (0.29) | 0.89 (0.55) | 1.67 (0.73) | 0.94 (0.90)
  Amplitude of WT daily rhythm at Morning condition | 1.00 (0.97) | 1.35 (0.47) | 1.45 (0.38) | 0.71 (0.68) | 0.73 (0.22) | 0.95 (0.67)
  Amplitude of WT daily rhythm at Night condition | 1.50 (0.83) | 1.05 (0.31) | 1.16 (0.33) | 0.54 (0.46) | 1.12 (0.26) | 0.86 (0.51)
  Amplitude of WT daily rhythm at Control condition | 1.83 (1.05) | 0.85 (0.56) | 1.51 (0.47) | 0.77 (0.34) | 0.95 (0.63) | 1.06 (0.97)

6. Secondary Outcome: Changes in Microbiota Diversity (Inverse Simpson Index)
Description: Microbiota diversity changes were measured using Inverse Simpson Index, accounting for both species richness (number of species) and evenness (distribution of species). A higher Inverse Simpson Index indicates greater diversity because it reduces the impact of dominant species and gives more weight to rarer species. Unlike the regular Simpson Index (which decreases as diversity increases), the inverse form is more intuitive: higher values mean a more diverse microbiota. This index is widely used in microbiome studies to compare microbial diversity across different samples, such as in health versus disease states.
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: Index
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 2 | 1 | 1 | 1 | 2
Index
  Inverse Simpson Index at Baseline | 39.72 (7.35) | 32.21 (11.26) | 25.37 (0) | 30.08 (0) | 52.15 (0) | 33.64 (22.46)
  Inverse Simpson Index Control condition | 30.31 (11.49) | 34.44 (3.81) | 37.38 (0) | 32.65 (0) | 41.94 (0) | 42.67 (1.39)
  Inverse Simpson Index Morning condition | 30.53 (19.08) | 29.60 (12.83) | 30.12 (0) | 18.70 (0) | 31.87 (0) | 34.49 (34.08)
  Evening condition | 28.70 (13.26) | 38.91 (3.75) | 37.73 (0) | 35.58 (0) | 28.25 (0) | 27.14 (19.15)

7. Secondary Outcome: Concentration of Total Short-chain Fatty Acids (SCFAs)
Description: Short-chain fatty acids (SCFAs) in fecal samples were analyzed using gas-liquid chromatography (GLC) with a GC-FID system. Samples were mixed with NaOH, lyophilized, and homogenized with formic acid, methanol, and an internal standard (2-ethyl butyric acid). After ultrasonic treatment and centrifugation, the supernatant was filtered and injected into an Agilent 7890A GC system equipped with a Nukol capillary column. Helium was used as the carrier gas, and the FID temperature was set at 220°C. SCFAs were identified by comparing retention times with authentic standards, and quantification was performed using calibration curves with a high correlation (R² = 0.99). Total average values of SCFA (acetate, propionate, other minorities) in each condition were calculated.
Time Frame: After 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: mmol/mg feces
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 2 | 3 | 1 | 1 | 1 | 1
mmol/mg feces
  Total SCFA Control condition | 419.93 (160.81) | 293.15 (107.81) | 588.49 (0) | 196.93 (0) | 659.92 (0) | 596.45 (0)
  Total SCFA Morning condition | 533.10 (171.38) | 450.68 (209.02) | 482.40 (0) | 876.56 (0) | 608.80 (0) | 426.75 (0)
  Total SCFA Evening condition | 377.78 (152.54) | 661.70 (217.39) | 552.32 (0) | 754.51 (0) | 890.21 (0) | 580.86 (0)

8. Secondary Outcome: Energy Intake
Description: The investigators will measure changes in total energy intake measured as kilocalories between baseline and after 2 weeks in each condition (no chocolate, Morning Chocolate, Night Chocolate) At baseline and during the 2 weeks of each condition, time-stamped photographs were captured with a cell phone app. Total energy intake during the 14 days of each condition was analyzed with the nutritional evaluation software (Grunumur 2.0 8).
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 3 | 3
kcal
  Energy intake at Baseline | 1177.20 (402.25) | 1987.20 (404.29) | 1558.15 (271.12) | 2044.61 (0) | 1843.39 (208.39) | 2031.93 (271.14)
  Energy intake at Morning condition | 1596.74 (340.18) | 2214.31 (122.01) | 2374.69 (248.37) | 2034.83 (0) | 1933.39 (109.42) | 2248.11 (220.18)
  Energy intake at Night condition | 1929.59 (295.25) | 2225.40 (26.95) | 2237.69 (570.40) | 2487.92 (0) | 2248.46 (64.52) | 2448.73 (589.64)
  Energy intake at Control condition | 1797.58 (431.61) | 1843.50 (405.89) | 2173.95 (722.95) | 1882.36 (0) | 1548.47 (97.43) | 1766.66 (358.91)

9. Secondary Outcome: Macronutrient Composition
Description: The investigators will measure macronutrient composition measured as and grams per day between baseline and after 2 weeks in each condition (no chocolate, Morning Chocolate, Night Chocolate). At baseline and during the 2 weeks of each condition, time-stamped photographs were captured with a cell phone app. Macronutrient composition during the 14 days of each condition was analyzed with the nutritional evaluation software (Grunumur 2.0 8).
Time Frame: Baseline and after 2 weeks in each condition
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Morning Chocolate, Then Evening/Night Chocolate and Control Chocolate | Morning Chocolate, Then Control Chocolate and Evening/Night Chocolate | Evening/Night Chocolate, Then Morning Chocolate and Control Chocolate | Evening/Night Chocolate, Then Control Chocolate and Morning Chocolate | Control Chocolate, Then Morning Chocolate and Evening/Night Chocolate | Control Chocolate, Then Evening/Night Chocolate and Morning Chocolate
Number analyzed (Participants) | 3 | 3 | 5 | 1 | 3 | 3
grams/day
  Carbohydrates at Baseline | 111.39 (45.57) | 198.72 (30.66) | 182.84 (45.09) | 202.74 (0) | 164.86 (40.63) | 171.72 (39.89)
  Fat at Baseline | 58.78 (13.50) | 101.32 (28.72) | 66.44 (19.62) | 103.12 (0) | 92.87 (10.77) | 116.83 (15.56)
  Protein at Baseline | 45.56 (10.26) | 76.59 (10.76) | 58.37 (17.75) | 75.46 (0) | 75.28 (6.49) | 71.53 (11.08)
  Carbohydrates at Morning condition | 156.78 (21.09) | 256.53 (36.88) | 239.23 (39.60) | 214.30 (0) | 174.29 (31.04) | 217.07 (29.02)
  Fat at Morning condition | 76.97 (19.28) | 102.66 (14.92) | 122.65 (14.30) | 99.44 (0) | 103.31 (19.58) | 119.00 (9.83)
  Protein at Morning condition | 67.17 (15.70) | 74.10 (6.43) | 80.39 (10.18) | 66.61 (0) | 70.88 (2.34) | 83.28 (7.52)
  Carbohydrates at Night condition | 174.53 (21.70) | 237.02 (10.58) | 232.31 (50.15) | 233.36 (0) | 207.00 (27.04) | 233.52 (76.51)
  Fat at Night condition | 102.36 (21.85) | 109.84 (2.46) | 112.92 (34.86) | 139.51 (0) | 115.74 (7.39) | 131.45 (25.01)
  Protein at Night condition | 75.34 (10.11) | 76.99 (5.70) | 76.04 (20.96) | 71.53 (0) | 76.30 (9.20) | 87.47 (21.96)
  Carbohydrates at Control condition | 141.53 (30.34) | 212.31 (91.16) | 218.36 (76.08) | 179.15 (0) | 137.00 (43.42) | 166.02 (28.94)
  Fat at Control condition | 97.20 (32.61) | 80.99 (8.32) | 110.66 (39.32) | 97.12 (0) | 76.80 (12.32) | 90.09 (25.22)
  Protein at Control condition | 75.15 (19.68) | 68.27 (16.37) | 78.30 (22.18) | 70.04 (0) | 65.44 (10.44) | 70.04 (10.08)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for each arm in the three conditions (Morning, Evening/Night, Control) during two weeks each, along with washout periods of one week between conditions. In total, adverse events were reported for up to eight weeks.
Groups:
- Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Morning Condition; Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Evening Condition; Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Evening/Night Chocolate and Control Chocolate: Behavioral: Evening/Night Chocolate Eating 100gr of milk chocolate within (1 hours of habitual bedtime) Behavioral: Control Chocolate Eating no milk chocolate or other chocolate
- Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Morning Condition; Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Evening Condition; Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Control Chocolate and Evening/Night Chocolate: Behavioral: Control Chocolate Eating no milk chocolate or other chocolate Behavioral: Evening/Night Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual bedtime)
- Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Morning Condition; Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Evening Condition; Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Morning Chocolate and Control Chocolate: Behavioral: Morning Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual waketime) Behavioral: Control Chocolate Eating no milk chocolate or other chocolate
- Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Morning Condition; Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Evening Condition; Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Control Chocolate and Morning Chocolate: Behavioral: Control Chocolate Eating no milk chocolate or other chocolate. Behavioral: Morning Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual waketime)
- Control Chocolate First, Second Morning Chocolate and Evening/Night Chocolate: Morning Condition; Control Chocolate First, Then Morning Chocolate and Evening/Night Chocolate: Evening Condition; Control Chocolate First, Second Morning Chocolate and Evening/Night Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Morning Chocolate and Evening/Night Chocolate: Behavioral: Morning Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual waketime) Behavioral: Evening/Night Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual bedtime)
- Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Morning Condition; Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Evening Condition; Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Control Condition: The intervention is eating chocolate within one hour of habitual waketime.
  Evening/Night Chocolate and Morning Chocolate: Behavioral: Evening/Night Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual bedtime) Behavioral: Morning Chocolate Eating 100gr of milk chocolate (within 1 hours of habitual waketime)
Arm/Group | Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Morning Condition | Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Morning Condition | Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Morning Condition | Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Morning Condition | Control Chocolate First, Second Morning Chocolate and Evening/Night Chocolate: Morning Condition | Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Morning Condition | Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Evening Condition | Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Evening Condition | Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Evening Condition | Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Evening Condition | Control Chocolate First, Then Morning Chocolate and Evening/Night Chocolate: Evening Condition | Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Evening Condition | Morning Chocolate First, Second Evening/Night Chocolate and Control Chocolate: Control Condition | Morning Chocolate First, Second Control Chocolate and Evening/Night Chocolate: Control Condition | Evening/Night Chocolate First, Second Morning Chocolate and Control Chocolate: Control Condition | Evening/Night Chocolate First, Second Control Chocolate and Morning Chocolate: Control Condition | Control Chocolate First, Second Morning Chocolate and Evening/Night Chocolate: Control Condition | Control Chocolate First, Second Evening/Night Chocolate and Morning Chocolate: Control Condition
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3 | 0/3 | 0/3 | 0/5 | 0/2 | 0/3 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes